CLINICAL TRIAL: NCT04013399
Title: Obstructive Sleep Apnea Treatment and Insulin Sensitivity in Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed due to Covid-19
Sponsor: Barnes-Jewish Hospital (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Sarah Farabi, Assistant Professor, Barnes-Jewish Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201905166
Record Dates: First submitted 2019-05-23; First posted 2019-07-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Obstructive Sleep Apnea; Pregnancy Related; Insulin Sensitivity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Insulin Resistance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Positive Airway Pressure (Experimental): Women will receive Continuous Positive Airway Pressure (CPAP) for one month.
  Interventions: Device: Continuous Positive Airway Pressure
- Control (No Intervention): Women will receive standard prenatal care.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — The device is an auto-adjusting pressure device with an integrated humidifier. Pressure is adjusted based on airway resistance.
  Arms: Continuous Positive Airway Pressure

SUMMARY:
This study will evaluate the effect of treatment of obstructive sleep apnea on insulin sensitivity in pregnant women. Women in their third trimester of pregnancy will be randomized to receive treatment or no treatment for one month.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) worsens over pregnancy and is related to increased risk of gestational diabetes. Despite the fact that sleep disturbances are common during pregnancy, OSA remains under-diagnosed, and poorly understood particularly in pregnancies affected by obesity. At least 25 percent of pregnancies are now affected by obesity, a leading risk factor for OSA, yet the effect of treatment of OSA on patterns of metabolic function and specifically decreased insulin sensitivity in pregnant women with obesity is a neglected area with major therapeutic implications to improve maternal health. Inflammation with OSA may decrease insulin sensitivity. Continuous positive airway pressure (CPAP) is a known effective treatment for OSA and has been shown to improve insulin sensitivity outside of pregnancy. Our overall hypothesis is that, compared with standard care, CPAP will improve nighttime breathing, blood and tissue oxygenation, decrease markers of inflammation, and increase insulin sensitivity. Using a randomized controlled trial, we will determine the effect of CPAP on metabolic dysfunction induced by OSA in pregnant women with obesity.

ELIGIBILITY:
Inclusion Criteria:

* 28-32 weeks pregnant
* Age 20-39
* BMI 30-40 kg/m2 pre-pregnancy (or first trimester)
* Obstructive Sleep Apnea (AHI≥15)
* Have a singleton pregnancy

Exclusion Criteria:

* Diabetes (GDM, type 1 or type 2)
* Using beta blockers or glucocorticoids
* Have children who are ≤2 yrs old (risk of disrupted sleep)
* Diagnosed sleep disorders (other than sleep apnea)
* Night work schedule
* Diagnosed congestive heart failure
* Diagnosed lung disease (e.g. asthma, chronic obstructive pulmonary disease)
* Pre-gestational hypertension

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Degree of Insulin Sensitivity measured by Matsuda Index by Oral glucose Tolerance Test | 1 month
  Change in whole body insulin sensitivity measured using Matsuda Index
Percent of Oxygen in blood by pulse oximetry | 1 month
  Change in oxygen saturation measured by pulse oximetry

SECONDARY OUTCOMES:
Percent of Oxygen in Adipose Tissue measured by oxygen tension probe | 1 month
  Change in adipose tissue oxygenation measured by oxygen tension
Concentration of inflammatory gene expression in adipose Tissue measured by RNA and DNA sequencing | 1 month
  Change in adipose tissue gene expression of inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No